CLINICAL TRIAL: NCT01171820
Title: SPIRIT V: A Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: SPIRIT V: A Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Patients With de Novo Coronary Artery Lesions (Diabetic Sub-Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-369 Diabetic Sub-study
Record Dates: First submitted 2010-04-01; First posted 2010-07-29 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; Angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAXUS® Liberté™ (Active Comparator)
  Interventions: Device: TAXUS® Liberté™
- XIENCE V® EECSS (Active Comparator)
  Interventions: Device: XIENCE V® EECSS

INTERVENTIONS:
Device: TAXUS® Liberté™ — Drug eluting stent implantation stent in the treatment of coronary artery disease in participants with Diabetes
  Arms: TAXUS® Liberté™
Device: XIENCE V® EECSS — Drug eluting stent implantation stent in the treatment of coronary artery disease in participants with Diabetes
  Arms: XIENCE V® EECSS

SUMMARY:
The purpose of this Clinical Evaluation is a continuation in the assessment of the performance of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in the treatment of patients with de novo coronary artery lesions in patients (Diabetic sub-study).

DETAILED DESCRIPTION:
The SPIRIT V Clinical Evaluation consists of two concurrent studies,the Diabetic sub-study and the Registry.

The SPIRIT V Diabetic sub-study is a prospective, randomized, active-controlled, single blind, parallel two-arm multi-center study comparing the XIENCE V® EECSS to the TAXUS® Liberté™ in the treatment of diabetic patients with coronary artery lesions who will fulfill the eligibility criteria. Approximately 300 patients will be randomized (2:1) against the TAXUS® Liberté™ coronary stent system. These patients will be recruited in up to 40 selected sites.

The long term safety and efficacy of the XIENCE V EECSS have been demonstrated in the SPIRIT FIRST trial up to 5 years, the SPIRIT II trial up to 4 years, and in the SPIRIT III Randomized Control Trial (RCT) up to 3 years. In addition, these pre-approval studies have shown low rates of Target Vessel Failure and Major Adverse Cardiac Events (MACE) that were observed to plateau or gradually decline after about 1 year and were consistently lower than the comparator arm of each study. This benefit in MACE is sustained for up to 5 years and is also independent of the first year results.

The post approval SPIRIT V study demonstrated that the use of the XIENCE EECSS in complex lesions in a real-world population resulted in 1 year MACE, Stent Thrombosis and Target Lesion Revascularization rates that are comparable to those of the previously mentioned pre-approval studies which included patients with more restricted inclusion / exclusion criteria.

Therefore, based on existing data from these trials, Abbott Vascular has decided to discontinue further follow up in the SPIRIT V Diabetic study after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the XIENCE V® EECSS and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site
* diagnosed with diabetes, as documented by medical history.
* evidence of myocardial ischemia
* acceptable candidate for coronary artery bypass grafting (CABG) surgery
* agree to undergo all clinical investigation plan (CIP)-required follow-up examinations
* artery morphology and disease is suitable to be optimally treated with a maximum of 4 planned stents
* maximum of one, de novo, target lesion per native major epicardial vessel or side branch
* target vessel reference diameter must be between 2.25 mm and 4.0 mm by visual estimate
* target lesion ≤ 28 mm in length by visual estimate
* target lesion must be in a major artery or branch with a visually estimated stenosis of > 50% and < 100% and a TIMI flow > 1

Exclusion Criteria:

* known diagnosis of acute myocardial infarction within 72 hours preceding the index procedure
* current unstable arrhythmias
* Left ventricular ejection fraction < 30%
* received a heart or any other organ transplant or is on a waiting list for any organ transplant
* receiving or scheduled to receive chemotherapy or radiation therapy within 30 days prior to or after the procedure.
* receiving immunosuppression therapy or has known immunosuppressive or autoimmune disease
* known hypersensitivity or contraindication to specific agents
* elective surgery is planned within the first 9 months after the procedure that will require discontinuing either aspirin or clopidogrel
* platelet count limits, white blood cell limits or documented or suspected liver disease
* renal insufficiency
* history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Cerebrovascular accident or transient ischemic attack within the past 6 months
* significant GI or urinary bleed within the past 6 months
* history of other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse that may cause non-compliance with the CIP, confound the data interpretation or is associated with a limited life expectancy (i.e. less than one year)

Target lesion meets any of the following criteria:

* In-stent restenotic
* aorto-ostial location (within 3 mm)
* left main location
* located within 2 mm of the origin of the left anterior descending artery (LAD) or left circumflex artery (LCX)
* located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft (defined as vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation)
* lesion involving a side branch ≥ 2.5 mm in diameter
* lesion involving a side branch with > 50% stenosis by visual estimation Lesion involving a side branch requiring predilatation
* located in a major epicardial vessel that has been previously treated with brachytherapy
* located in a major epicardial vessel or a side branch that has been previously treated with any type of percutaneous intervention (e.g., balloon angioplasty, cutting balloon, atherectomy), < 9 months prior to the index procedure
* total occlusion (TIMI flow 0), prior to wire crossing
* excessive tortuosity proximal to or within the lesion
* extreme angulation (≥ 90%) proximal to or within the lesion
* heavy calcification

The target vessel contains visible thrombus

Patient has a high probability that a procedure other than pre-dilatation, stenting and post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. brachytherapy)

Patient has additional clinically significant lesion(s) (> 50% diameter stenosis) in a target vessel or side branch for which an intervention within 9 months after the index procedure may be required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, MD, Principal Investigator — International Heart Center Rhein-Ruhr, Essen, Germany; Upendra Kaul, MD, Principal Investigator — Fortis Hospital, New Delhi, India
Locations (28):
- Salzburger Landeskliniken, Salzburg, Austria
- France (2):
  - C.H.U. - Hopital Michallon, Grenoble
  - CHU Lille - Hôpital Cardiologique, Lille
- Germany (4):
  - Herzzentrum, Bernau
  - Universitätsklinikum, Heidelberg
  - Lukas Krankenhaus Neuss, Neuss
  - Herzzentrum Siegburg GmbH, Siegburg
- Sheba Medical Center, Ramat Gan, Israel
- Italy (5):
  - Azienda Ospedaliera Riuniti, Bergamo
  - Ospedale Civile, Mirano
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera S. Gdi Dio Salerno, Salerno
- Institute Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Medisch Centrum Alkmaar, Alkmaar
  - Maasstad Ziekenhuis, Rotterdam
- Medical University of Bydgoszcz, Bydgoszcz, Poland
- Spain (8):
  - General De Alicante, Alicante
  - Hospital Belvigte de Barcelona, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Clinico San Carlos, Madrid
  - Hospital Puerta de Hierro, Madrid
  - La Paz, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital General de Valencia, Valencia
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand
- United Kingdom (2):
  - Wessex Cardiac Unit, Southampton, Southampton
  - King's College Hospital, London

REFERENCES:
- See also: SPIRIT V registry arm — http://clinicaltrials.gov/ct2/show/NCT00402272?term=SPIRIT+V&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 324 subjects were recruited at 32 sites. Eligible subjects invited to participate, in-hospital or in-clinic and required to provide signed informed consent prior to enrollment. Final eligibility based on angiographic inclusion criteria prior to the intended procedure. Dates of recruitment: April 28, 2007 to October 6, 2008.
Pre-assignment Details: Subjects were randomized via telephone randomization and stratified by insulin treatment status, number of lesions treated-single vs. multiple. Randomization only occurred after verification of the inclusion/exclusion criteria and successful pre-dilatation. See the Eligibility Criteria (inclusion/exclusion criteria) for details.
Groups:
- TAXUS® Liberté™: Patients receiving the TAXUS® Liberté™ stent during PCI
- XIENCE V® EECSS: Patients receiving the XIENCE V® EECSS stent during percutaneous coronary intervention (PCI)
Period: Overall Study
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Started | 106 | 218
Completed | 100 | 212
Not Completed | 6 | 6
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — 1-Year Missed Visit | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- XIENCE V® EECSS: Patients receiving the XIENCE V® EECSS stent during PCI
- Total: Total of all reporting groups
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS | Total
Number analyzed (Participants) | 106 | 218 | 324
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 102 | 151
  >=65 years | 57 | 116 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.75 (8.95) | 65.32 (9.61) | 65.46 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 66 | 101
  Male | 71 | 152 | 223
Region of Enrollment [Number; unit: participants]
  France | 2 | 7 | 9
  Thailand | 0 | 2 | 2
  Spain | 57 | 87 | 144
  Poland | 8 | 17 | 25
  Malaysia | 1 | 13 | 14
  Austria | 2 | 8 | 10
  Israel | 1 | 1 | 2
  Netherlands | 1 | 12 | 13
  Germany | 14 | 22 | 36
  United Kingdom | 3 | 6 | 9
  Italy | 17 | 43 | 60

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Loss (LL)
Description: In-stent minimal lumen diameter (MLD) post-procedure minus (-) in-stent MLD at follow-up
Time Frame: 270 days
Population: Analysis based on intention to treat (ITT) population. Patients were required to have angiographic follow-up to provide this endpoint information. Some patients not completing the study, did not have this follow up.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 110 | 249
millimeters | 0.39 (0.49) | 0.19 (0.37)

2. Secondary Outcome: Clinical Device Success (Per-lesion)
Description: Successful delivery and deployment of the study stent (in overlapping stent setting a successful delivery and deployment of the first and second study stent) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of final residual stenosis of less than 50% of the target lesion by quantitative coronary angiography (QCA) (by visual estimation if QCA unavailable), without use of a device outside the assigned treatment strategy.
Time Frame: immediately post-procedure
Population: Analysis based on intention to treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (Lesions) | 133 | 289
Percentage of lesions | 98.50 [94.67 to 99.82] | 97.58 [95.07 to 99.02]

3. Secondary Outcome: Clinical Procedure Success (Per-patient)
Description: Successful delivery and deployment of the study stent or stents at the intended target lesion and successful withdrawal of the stent delivery system with attainment of final residual stenosis of less than 50% of the target lesion by quantitative coronary angiography (QCA) (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of cardiac death, MI attributed to the target vessel and/or CI-TLR during the hospital stay with a maximum of first seven days post index procedure. In multiple lesion setting each lesion must meet clinical procedure success.
Time Frame: immediately post-procedure
Population: The sample size for clinical procedure success is based on the number of evaluable patients, for whom data is available to define clinical procedure success.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 102 | 212
Percentage of participants | 93.14 [86.37 to 97.20] | 96.70 [93.32 to 98.66]

4. Secondary Outcome: In-segment Late Loss
Description: In-segment minimal lumen diameter (MLD) post-procedure minus (-) in segment MLD at follow-up
Time Frame: 270 days
Population: Analysis based on intention to treat (ITT) population. Patients were required to have angiographic follow-up to provide this endpoint information. Some patients not completing the study, did not have this follow up. The number of analyzed represents number of patients randomized.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 109 | 249
millimeters | 0.22 (0.45) | 0.12 (0.42)

5. Secondary Outcome: Proximal Late Loss
Description: Proximal Minimum Lumen Diameter (MLD) post-procedure minus proximal MLD at follow-up
Time Frame: 270 day
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 104 | 241
millimeters | 0.17 (0.33) | 0.13 (0.39)

6. Secondary Outcome: Distal Late Loss
Description: Distal Minimum Lumen Diameter (MLD) post-procedure minus distal MLD at follow-up
Time Frame: 270 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 107 | 247
millimeters | 0.0 (0.34) | 0.0 (0.3)

7. Secondary Outcome: In-stent Angiographic Binary Restenosis Rate
Description: Percent of patients with a follow-up percent diameter stenosis of ≥ 50% per QCA.
Time Frame: 270 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 115 | 261
Percentage of participants | 6.1 [2.48 to 12.14] | 3.1 [1.33 to 5.95]

8. Secondary Outcome: In-segment Angiographic Binary Restenosis Rate
Description: Percent of patients with a follow-up percent diameter stenosis of ≥ 50% per QCA.
Time Frame: 270 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 110 | 255
Percentage of participants | 6.4 [2.60 to 12.67] | 7.5 [4.55 to 11.39]

9. Secondary Outcome: In-stent Percent Diameter Stenosis (% DS)
Description: This number represents the average of percent diameter stenosis found on examination of all the lesions analyzed.
  This value calculated as 100 * (1 - minimum lumen diameter/reference vessel diameter) (MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: 270 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent diameter stenosis
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 115 | 261
Percent diameter stenosis | 20.70 (16.02) | 14.33 (13.34)

10. Secondary Outcome: In-segment Percent Diameter Stenosis (% DS)
Description: This number represents the average of percent diameter stenosis found on examination of all the lesions analyzed.
  This value calculated as 100 * (1 - MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: 270 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent diameter stenosis
Units Other Than Participants: lesions
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Number analyzed (lesions) | 110 | 255
Percent diameter stenosis | 23.87 (15.25) | 22.42 (15.05)

11. Secondary Outcome: Adjudicated Stent Thrombosis (Confirmed/Definite, Probable, Possible)
Description: The Clinical Event Committee will adjudicate the events according to the definitions developed by the Academic Research Consortium (ARC), as published in Circulation (Cutlip, D.E., et al., Clinical End Points in Coronary Stent Trials: A Case for Standardized Definitions. Circulation, 2007. 115: p. 2344-2351.)
  Stent thrombosis was defined according to the ARC guidelines as follows: definite: acute coronary syndrome and angiographic or pathological confirmation of stent thrombosis; probable: unexplained death ≤30 days or any MI that is related to acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis; and possible: unexplained death >30 days after stent placement.
Time Frame: 0 to 37 days
Population: Analysis based on intention to treat (ITT) population. The number of patients analyzed excludes subjects who were lost-to-follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Percentage of participants | 0.94 [0.02 to 5.14] | 0.00 [0.00 to 1.68]

12. Secondary Outcome: Adjudicated Stent Thrombosis (Confirmed/Definite, Probable, Possible)
Description: as for outcome 11
Time Frame: 254 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 217
Percentage of participants | 2.83 [0.59 to 8.05] | 0.46 [0.01 to 2.54]

13. Secondary Outcome: Adjudicated Stent Thrombosis (Confirmed/Definite, Probable, Possible)
Description: as for outcome 11
Time Frame: 365 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 104 | 215
Percentage of participants | 2.88 [0.60 to 8.20] | 0.47 [0.01 to 2.56]

14. Secondary Outcome: Adjudicated Revascularizations (Target Lesion Revascularization (TLR)/ Target Vessel Revascularization (TVR)/Any Revascularization) Both Clinically-indicated and Not Clinically-indicated.
Description: TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion was defined as the treated segment from 5 mm proximal and 5 mm distal to the stent.
  TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel was defined as the entire major coronary vessel proximal and distal to the target lesion, including upstream and downstream branches and the target lesion itself.
  A revascularization is considered clinically indicated if angiography at follow-up shows a %DS ≥ 50% and if one of the following occurs: history of recurrent angina pectoris due to the target vessel; signs of ischemia at rest or during exercise test due to target vessel; abnormal results of any invasive diagnostic test; TLR or TVR with a % DS ≥ 70% even in the absence of the above mentioned ischemic signs.
Time Frame: 37 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Percentage of participants | 2.83 [0.59 to 8.05] | 1.38 [0.28 to 3.97]

15. Secondary Outcome: Adjudicated Revascularizations (Target Lesion Revascularization (TLR)/ Target Vessel Revascularization (TVR)/Any Revascularization) Both Clinically-indicated and Not Clinically-indicated.
Description: as for outcome 14
Time Frame: 254 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 217
Percentage of participants | 4.72 [1.55 to 10.67] | 6.45 [3.57 to 10.59]

16. Secondary Outcome: Adjudicated Revascularizations (Target Lesion Revascularization (TLR)/ Target Vessel Revascularization (TVR)/Any Revascularization) Both Clinically-indicated and Not Clinically-indicated.
Description: as for outcome 14
Time Frame: 393 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 104 | 215
Percentage of participants | 14.42 [8.30 to 22.67] | 20.93 [15.70 to 26.99]

17. Secondary Outcome: Adjudicated Composite Endpoint of Cardiac Death, Myocardial Infarction (MI) Attributed to the Target Vessel and Clinical-indicated Target Lesion Revascularization (CI-TLR)
Description: Cardiac death: Any death due to proximate cardiac cause (eg, myocardial infarction, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure related deaths, including those related to concomitant treatment, will be classified as cardiac death.
  MI- due to target vessel: All infarcts that cannot be clearly attributed to a vessel other than the target vessel will be considered related to the target vessel.
  Clinical-indicated Target Lesion Revascularization (CI-TLR): TLR with evidence of diameter stenosis ≥ 50% determined by QCA; or in the case of any one of the following: new recurrent history of angina pectoris, ischemic signs, abnormal results in diagnostic tests, or TLR >=70% in the absence of the above signs.
Time Frame: 37 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Percentage of participants | 7.55 [3.31 to 14.33] | 2.29 [0.75 to 5.27]

18. Secondary Outcome: Adjudicated Composite Endpoint of Cardiac Death, Myocardial Infarction (MI) Attributed to the Target Vessel and Clinical-indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 17
Time Frame: 254 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 217
Percentage of participants | 9.43 [4.62 to 16.67] | 5.53 [2.89 to 9.46]

19. Secondary Outcome: Adjudicated Composite Endpoint of Cardiac Death, Myocardial Infarction (MI) Attributed to the Target Vessel and Clinical-indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 17
Time Frame: 393 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 104 | 215
Percentage of participants | 12.50 [6.83 to 20.43] | 11.16 [7.28 to 16.15]

20. Secondary Outcome: Adjudicated Composite Endpoint of All Death, MI and Target Vessel Revascularization (TVR)
Description: Death defined by the Academic Research Consortium is as follows: All death is considered to be cardiac death unless an unequivocal noncardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal noncardiac disease (eg, cancer, infection) should be classified as cardiac.
  Myocardial infarction: Myocardial Infarction Classification and Criteria for Diagnosis as defined by the Academic Research Consortium.
  Target Vessel Revascularization (TVR): Target vessel revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
Time Frame: 37 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Percentage of participants | 8.49 [3.96 to 15.51] | 2.29 [0.75 to 5.27]

21. Secondary Outcome: Adjudicated Composite Endpoint of All Death, MI and Target Vessel Revascularization (TVR)
Description: as for outcome 20
Time Frame: 254 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 217
Percentage of participants | 11.32 [5.99 to 18.94] | 6.45 [3.57 to 10.59]

22. Secondary Outcome: Adjudicated Composite Endpoint of All Death, MI and Target Vessel Revascularization (TVR)
Description: as for outcome 20
Time Frame: 393 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 104 | 215
Percentage of participants | 16.35 [9.82 to 24.88] | 16.28 [11.61 to 21.91]

23. Secondary Outcome: Adjudicated Composite Endpoint of All Death, Any Myocardial Infarction (MI) and Any Revascularization (TLR/TVR/Non-TVR)
Description: Death defined by the Academic Research Consortium is as follows: All death is considered to be cardiac death unless an unequivocal noncardiac cause can be established.
  MI- due to target vessel: All infarcts that cannot be clearly attributed to a vessel other than the target vessel will be considered related to the target vessel.
  Any revascularization: TLR or TVR or non-TVR
Time Frame: 37 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 218
Percentage of participants | 10.38 [5.30 to 17.81] | 3.21 [1.30 to 6.50]

24. Secondary Outcome: Adjudicated Composite Endpoint of All Death, Any Myocardial Infarction (MI) and Any Revascularization (TLR/TVR/Non TVR)
Description: as for outcome 23
Time Frame: 254 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 106 | 217
Percentage of participants | 14.15 [8.14 to 22.26] | 9.68 [6.09 to 14.41]

25. Secondary Outcome: Adjudicated Composite Endpoint of All Death, Any Myocardial Infarction (MI) and Any Revascularization (TLR/TVR/Non TVR)
Description: as for outcome 23
Time Frame: 393 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Number analyzed (Participants) | 104 | 215
Percentage of participants | 23.08 [15.38 to 32.36] | 24.19 [18.62 to 30.48]

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were 324 (218 XV, 106 TX) total patients in the dataset. To qualify as an At-Risk patient, the patient must have completed the study AND/OR have at least one adverse event. Applying this rule, the At-Risk population therefore totaled 215 XV and 105 TX and is not equal to the number of patients enrolled.
Arm/Group | TAXUS® Liberté™ | XIENCE V® EECSS
Serious Adverse Events (participants affected / at risk) | 41/105 | 100/215
Other Adverse Events (participants affected / at risk) | 13/105 | 26/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS® Liberté™ (N=105) | XIENCE V® EECSS (N=215)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Angina pectoris (Cardiac disorders) | 13 (14) | 25 (29)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery restenosis (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 13 (13)
In-stent coronary artery restenosis (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 9 (9) | 6 (8)
Myocardial infarction, acute (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 4 (4)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (4)
Noncardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Instent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 2 (2)
Ejection fraction decreased (Investigations) | 2 (2) | 0 (0)
Troponin T (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Diabetic foot (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meniscus lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkins disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip andor oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 4 (5)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 2 (2)
Diabetes mellitus management (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 3 (4)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Retroperitoneal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS® Liberté™ (N=105) | XIENCE V® EECSS (N=215)
Angina pectoris (Cardiac disorders) | 12 (13) | 14 (14)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less